CLINICAL TRIAL: NCT05179915
Title: The Effect of Sacral Region-focused Therapeutic Touch Applied During the Latent Phase of Labour on Hormone Levels, Labour Comfort and Perception: A Randomized Sham Controlled Trialt
Brief Title: Effect of Therapeutic Touch on Labor Pain and Hormone Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ebru Gözüyeşil, Associate Prof., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: egozuyesil@cu.edu.tr
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-02

CONDITIONS: Therapeutic Touch; Childbirth
Keywords: Labor Pain; Therapeutic Touch; Childbirth; Hormones
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: A randomized sham controlled trial design was used in the study, which was conducted with 50 primiparous pregnant women. While Therapeutic Touch (25) focused on sacral region was applied in the intervention group, Sham Therapeutic Touch (25) was applied in the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to ensuring the blinding of the participants in the study, blinding was also performed during the data collection, hormone values analysis, statistics and reporting stages. Women who agreed to participate in the study were not informed about the group they were assigned to. Since the participants did not know to which group they were assigned, the study was conducted in a single-blind design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be administered 15-minute therapeutic touch focused on sacral region the latent phase and after it finishes, the participating pregnant woman will be asked to rest for 30 minutes.
  Interventions: Other: Therapeutic Touch focused on sacral region
- Placebo Group (Placebo Comparator): After the mimic (sham) therapeutic touch focused on sacral region , the pregnant woman will be asked to rest for 30 minutes.
  Interventions: Other: Therapeutic Touch focused on sacral region

INTERVENTIONS:
Other: Therapeutic Touch focused on sacral region — In the latent phase of labor, the field energy of the sacral region will be cleared for an average of 15 minutes.
  Other Names: Placebo Touch (Mimic Touch) focused on sacral region

SUMMARY:
This study was conducted to determine the effect of sacral region-focused therapeutic touch applied during the latent phase of labour on hormone levels, labour comfort, and perception.

A randomized sham controlled trial design was used in the study, which was conducted with 50 primiparous pregnant women. While Therapeutic Touch (25) focused on sacral region was applied in the intervention group, Sham Therapeutic Touch (25) was applied in the control group. Data were collected using a Personal Information Form, the Visual Analogue Scale, a Hormone Values Follow-up Form, the Childbirth Comfort Questionnaire and the Perception of Birth Scale.

Keywords: Labor Pain,Therapeutic Touch, Childbirth, Hormones

DETAILED DESCRIPTION:
Aim: This study was conducted to determine the effect of sacral region-focused therapeutic touch applied during the latent phase of labour on hormone levels, labour comfort, and perception.

Method: This randomised sham controlled experimental trial was conducted with two groups (intervention and control groups) in a state hospital between 08 March 2022 and 01 April 2023. The sample size of the study was calculated using the G*power 3.1.9.6 programme. As a result of the calculation, twenty-five pregnant women for each group were included in the study. While Therapeutic Touch (TT) focused on sacral region was applied in the intervention group, Sham Therapeutic Touch (STT) was applied in the control group. Data were collected using a Personal Information Form, the Visual Analogue Scale (VAS), a Hormone Values Follow-up Form, the Childbirth Comfort Questionnaire (CCQ) and the Perception of Birth Scale (PBS). IBM SPSS V25 programme was used for statistical analysis of the study. The statistical significance was assessed at the level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being primipara,
* Having a gestational age of 38-42 weeks,
* Planning to have a normal vaginal delivery,
* Having a 3-4 cm dilation in the latent phase,
* Having a single fetus and head presentation,
* Speaking and communicating in Turkish,
* Agreeing to participate in the study,
* Having no high-risk pregnancy.

Exclusion Criteria:

* Receiving induction,
* Receiving labor analgesia/anesthesia,
* Having sensitivity or problems with touch,
* Having to leave during the intervention due to some reasons such as medical procedures, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 50 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | VAS were evaluated after application 30 minutes in each groups.
  VAS is a one-dimensional scale that objectively assesses pregnant woman's perception of pain. VAS is a 100 mm scale (10-cm) that represents lack of pain (0=no pain) on one end and worst possible pain (10=severe pain) on the other end; the scale is used to determine the severity of pain quantitatively. The patient marks any point between the two ends that describe his/her pain severity. The point between lack of pain and the point indicated by the patient is measured using a ruler and recorded as cm. These numeric values indicate the pregnant woman's pain severity.

SECONDARY OUTCOMES:
The Perception of Birth Scale (PBS) | PBS were evaluated after delivery in each groups.
  MPLS PBS,is a measurement tool that assesses how mothers perceive their experiences in normal delivery or planned cesarean sections. The sub-scales of the scale include experiences during labor (7 items: 3, 5, 6, 8, 15, 17, 18), experiences during the pain phase of labor (7 items; 1, 2, 4, 7, 9, 10, 16), end of labor (4 items: 22, 23, 24, 25), partner involvement (4 items; 11,12,20,21), and awareness (3 items; 13,14,19). Each item in the MPLS is rated between 1 and 5: 1-Never, 2-A little, 3-Moderate, 4-A lot, and 5-Too much. Since Items 15-16-17-18-19 in the scale include negative statements, these items are scored reversely. Cronbach's alpha value of the scale was 0.90, and the alpha values obtained using two half-test methods were found 0.83 and 0.81.

OTHER OUTCOMES:
The Childbirth Comfort Questionnaire (CCQ) | CCQ were evaluated after application 30 minutes in each groups.
  The original name of the scale was the "Childbirth Comfort Questionnaire", and it was developed by Kerri Durnell Schuiling in 2003 based on Kolcaba's comfort theory (7). Turkish reliability and validity of the Childbirth Comfort Questionnaire were performed by Potur et al. (2015) (8). Cronbach's alpha coefficient of the scale was found 0.75. The 14-item scale is rated on a 5-point scale. Each item is responded considering the comfort in the delivery room. Each item in the original scale is reported to be scored between 1 and 5 (1=I strongly disagree, 2= I disagree, 3=I partly agree, 4= I agree, 5=I strongly agree). Scores to be obtained from the scale range between 14 and 70. Before the total score is calculated, item 2,4,6,9,12,13,14 should be reversed. While higher scores indicate a high level of comfort, lower scores indicate a low level of comfort.
Hormones | a maternal saliva sample for hormones was took pretest and posttest (after application in 30 minutes).
  Samples took from pregnant women two times for oxytocin, endorphin, and cortisol analyses, which will include right before starting Therapeutic Touch (TT) in the latent phase of the first phase of labor and 30 minutes after the therapeutic touch. The samples will be collected in 1.5 ml Eppendorf tubes that will have 70 μL spit sample. The samples will be taken to deep freezers at the Genetic Department of Medical Faculty at Çukurova University following the cold-chain rule and waited at -80 °C until the analysis day

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Gözüyeşil, PhD. Associate Professor,, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No